CLINICAL TRIAL: NCT05266157
Title: Lymphoedema and Nocturia/ Nocturnal Polyuria After Pelvic Lymph Node Dissection (LND) for Urogenital Cancer: Randomised Controlled Trial (Pilot)
Brief Title: Lymphoedema and Nocturia/ Nocturnal Polyuria After Pelvic Lymph Node Dissection for Urogenital Cancer
Acronym: UroLymph
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: s66072 RCT
Record Dates: First submitted 2022-01-17; First posted 2022-03-04 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Lower Limb Lymphedema; Urogenital Cancer
Keywords: manual lymph drainage
MeSH Terms: conditions — Urogenital Neoplasms | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Skin care, exercise and compression stocking:
  The patient has to wear custom-made compression thigh stocking(s) in case of unilateral/ bilateral swelling of the leg and has to wear a bermuda in case of swelling of the midline region. The patient continues the skin care and continues/ restarts exercise therapy with the home physical therapist 2 times a week. Frequency of exercises is gradually decreased: M1-3 2x/w, M4-6 1x/w, M7-9 1x/M; M10-12 only self-exercises.
  Interventions: Other: Usual care
- Additional manual lymph drainage (Experimental): Usual care + manual lymph drainage. Manual lymph drainage is performed by the home physical therapist. Every session lasts for 30 minutes.
  Frequency of manual lymph drainage is gradually decreased: M1-3 2x/w, M4-6 1x/w, M7-9 1x/M; M10-12 only self-MLD.
  Interventions: Other: Manual lymph drainage; Other: Usual care

INTERVENTIONS:
Other: Manual lymph drainage — Manual lymph drainage
  Arms: Additional manual lymph drainage
Other: Usual care — skin care, exercise and compression stocking

SUMMARY:
After the treatment of urogenital cancer, a person may develop lymphoedema of the leg(s) and/ or midline region. Lymphoedema is the result of a dysfunction in the lymphatic system and is characterized by excessive retention of lymphatic fluid in the interstitial compartment, adipose deposition and chronic tissue inflammation resulting in fibrosis. Clinical symptoms include abnormal tissue swelling, sensation of limb heaviness, erythema, pain, and impaired limb function.

The added value of manual lymph drainage, applied in patients with mild (early) lower limb lymphoedema and in addition to skin care, exercises and a compression stocking, has never been investigated.

Therefore, the objective of this randomised controlled pilot trial is to investigate the feasibility of a trial about the added value of manual lymph drainage (to skin care, exercises and wearing compression stocking) in patients with mild (early) lower limb lymphoedema. In fact, the investigators want to determine the sample size for a trial investigating the effectiveness of MLD and want to investigate the feasibility of the study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the prospective observational study and developing lymphoedema within the first year after surgery
* Before inclusion, written informed consent must be given according to ICH/GCP, and national/local regulations.

Inclusion criteria of the prospective observational study were:

* Non-metastatic urogenital cancer (i.e. prostate cancer or bladder cancer)
* Pelvic lymph node dissection

Exclusion Criteria: same as for the prospective observational study:

* Radiological evidence of metastatic disease based on pelvic CT/MRI and bone scan
* Clinical signs of chronic venous insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of lymphoedema-specific quality of life | Baseline-3-6-12 months
  Lymphoedema-specific quality of life will be evaluated using the Lymph-ICL-LL questionnaire: The Lymph-ICF-LL is a descriptive, evaluative tool containing 28 questions about impairments in function, activity limitations, and participation restrictions in patients with lower limb lymphoedema. The questionnaire has 5 domains: physical function, mental function, general tasks/household activities, mobility activities, and life domains/social life.
Change of volume of the lower limb | Baseline-3-6-12 months
  Volume measurements will be done at midline, leg and foot. Volume midline: circumference at the level of the hip and distance navel - pubic bone, with tapeline.
  Volume leg: circumference measurements in sitting position, with knee extension, foot supported by chair; reference point is the upper border of the patella and every 4cm up to the groin and to the ankle, with perimeter Volume foot: figure of 8 method: in sitting position, with knee extension, foot supported by chair and relaxed; with tapeline; make the figure 8 between the distal part of medial and lateral malleolus and the proximal border of metatarsal I and V
Change of health-related quality of life | Baseline-3-6-12 months
  Health-related quality of life will be assessed with the EuroQol EQ-5D-5L (questionnaire).
  The EQ-5D, developed by the EuroQol Group, is a generic HRQoL instrument commonly used for indirect utility measurement. It is a descriptive system for health states, encompassing 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), combined with a visual analogue scale ranging from "worst imaginable health state" to "best imaginable health state". Each health dimension has 5 levels of severity (EQ-5D-5L;5L: no problems, slight problems, moderate problems, severe problems,extreme problems /unable to).
  Each EQ-5D health state is labelled by a code, e.g. 21531, where each digit represents the severity level of a dimension. By convention, the order of dimensions is mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change of physical activity level | Baseline-3-6-12 months
  Physical activity will be assessed with the International Physical Activity Questionnaire (IPAQ).
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old.
Change of water content at the level of the legs/ midline region | Baseline-3-6-12 months
  Water content in the leg and midline region will be measured using the MoistureMeterD Compact.
Change of extracellular fluid at the level of the legs/ midline region | Baseline-3-6-12 months
  Extracellular fluid in the lower limb will be measured with bio-impedance spectroscopy.
Change of body weight | Baseline-3-6-12 months
  Body weight will be measured with an electronic balance
Infection rate | Baseline-6-12 months
  Number of infection episodes during the previous 6 months is questioned
Feasibility of the trial: number of patients accepting to participate | 12 months
  Number of patients accepting to participate in the randomized controlled pilot trial
Feasibility of the trial: information about the intervention | 12 months
  If the participant is randomised to the intervention group with manual lymph drainage, information is collected regarding the type of lymph drainage, the number of sessions and the duration of one session.
Feasibility of the trial: registration of difficulties | 12 months
  Difficulties concerning the intervention will be registered
Feasibility of the trial: Number of drop-outs in each group | 12 months
  The number of drop-outs in both the experimental as the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Flanders, Belgium